CLINICAL TRIAL: NCT01544751
Title: Metformin Versus Atorvastatin in Nonalcoholic Hepatic Steatosis: a Randomized Study
Brief Title: Nonalcoholic Fatty Liver Disease (NAFLD) Pharmacological Treatment: Metformin Versus Atorvastatin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prof Antonino Belfiore (Other)
Responsible Party: Sponsor-Investigator, Prof Antonino Belfiore, Full Professor, University Magna Graecia
Organization: University Magna Graecia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010.42
Record Dates: First submitted 2012-02-16; First posted 2012-03-06 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Nonalcoholic Fatty Liver Disease (NAFLD)
Keywords: NAFLD; metformin; atorvastatin; metabolic syndrome
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Metabolic Syndrome | interventions — Metformin; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low dose Metformin (Active Comparator): 500 mg twice a day for one year
  Interventions: Drug: Low dose metformin
- Metformin (Active Comparator): 1000 mg twice a day for one year
  Interventions: Drug: Metformin
- Atorvastatin (Active Comparator): 20 mg day
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Low dose metformin — 500 mg twice a day
  Arms: Low dose Metformin
Drug: Metformin — 1000 mg twice a day
  Arms: Metformin
Drug: Atorvastatin — 20 mg/day
  Arms: Atorvastatin

SUMMARY:
The first line approach to NAFLD is currently based on diet and lifestyle modification. Aim of our Unit is to compare the efficacy of two different doses of metformin (1 g/day and 2 g/day) with atorvastatin (20 mg/day) on amelioration of inflammatory and cardiometabolic parameters, ultrasound signs and clinical scores associated with liver fibrosis in early-stage NAFLD non-diabetic patients.

DETAILED DESCRIPTION:
Non alcoholic fatty liver disease (NAFLD) is a common liver disease that encompasses both simple steatosis and non alcoholic steatohepatitis (NASH.

There is currently no therapy that is of proven benefit for these liver disorders both of which are closely associated with insulin resistance and features of the metabolic syndrome such as obesity, hyperlipidaemia and type 2 diabetes mellitus. The first line approach to NAFLD is currently based on diet and lifestyle modification. However, dietary treatment is limited by the lack of compliance and the frequent regain of weight at follow-up.

Aim of our Unit is to compare the efficacy of two different doses of metformin (1 g/day and 2 g/day) with atorvastatin (20 mg/day) on amelioration of inflammatory and cardiometabolic parameters, ultrasound signs and clinical scores associated with liver fibrosis in early-stage NAFLD non-diabetic patients.

The investigators will enrol obese or overweight non-diabetic patients with ultrasonographic diagnosis of hepatic steatosis at early stage (NAFLD). The investigators will exclude from the study patients with clinical-biochemical and ultrasound markers of disease severity (age, BMI, lipid profile, AST, ALT, Angulo, BAAT and HAIR clinical fibrosis scores, signs of portal hypertension and posterior attenuation of the deep liver parenchyma at US). Patients who meet all eligibility criteria will be randomly assigned to one of three groups for 12 months of study treatment. The first group (n=50) will receive metformin (1g/day) plus dietary treatment; the second group (n=50) will be given metformin (2 g/day) and the third group (n=50) will be treated with atorvastatin (20 mg/day). All participants will be followed-up at 3, 6, 9, 12 months intervals after randomization. We will compare the effects of two doses of metformin with atorvastatin on the amelioration of both inflammatory (PCR, TNF-a , IL-6) and metabolic parameters (lipid profile, BMI, waist circumference, fasting glucose, 2-h glucose tolerance test, insulin, transaminases, adiponectin,leptin, HOMA-IR index and VAI index). Furthermore, we will assess the improvement under drug treatment of liver steatosis on the basis of US signs (liver echogenicity and stiffness) and of fibrosis scoring systems (Angulo, BAAT and HAIR scores).

In conclusion, considering the increasing prevalence of NAFLD and its strong association with cardiovascular diseases and cancer, the investigators expect to identify a safe pharmacological regimen that, in addition to dietary treatment, may ameliorate or even reverse this liver disease and the underlying risk factors. This study could have an important social impact in terms of both preventive and therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age <=55
* BMI <=40
* Total cholesterol <=280 mg/dl
* LDL <=180 mg/dl
* Triglycerides <=200 mg/dl
* AST and ALT in the normal range
* Signs of simple liver steatosis at ultrasonorography.

Exclusion criteria:

* Type 2 diabetes
* Heart disease
* Renal failure
* Smoking habit
* Alcohol intake of more than 20 g per day in the case of women and more than 30 g per day in the case of men
* Hepatic virus infection
* Autoimmune, metabolic or genetic liver diseases
* Use of drugs known to induce liver steatosis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-09; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with improvement of liver hyperechogenicity | one year
  We will investigate efficacy of metformin and atorvastatin in amelioration of liver hyperechogenicity and fibrosis scores.

SECONDARY OUTCOMES:
Number of Participants with amelioration of metabolic syndrome and HOMA-Index | one years
  We will investigate efficacy of metformin and atorvastatin in amelioration of metabolic parameters (change in the number of patients with metabolic syndrome from baseline and after treatment and amelioration of HOMA-Index from Baseline at one years).

CONTACTS AND LOCATIONS:
Overall Officials: Antonino Belfiore, Director, Study Director — Endocrinology Unit
Locations (1):
- Endocrinology Unit, Catanzaro, Catanzaro, Italy